CLINICAL TRIAL: NCT04696770
Title: Mindful Kangaroo Care: Mindfulness Intervention for Mothers During Skin-to-skin Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00089053
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Stress; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Intervention (Experimental): Four face-to-face direct coachings on Mindfulness technique at weekly intervals. The following will be the broad theme of each coaching session
  Week 1 - On the first encounter, the mothers will learn how to practice an introductory mindfulness technique to develop the awareness of any sensations felt in the body while holding their baby.
  Week 2 - On the second encounter, the mothers will learn how to practice a second mindfulness technique to create positive feelings in the body while holding their baby.
  During the third and fourth weekly encounters, the mothers will have a chance to ask their questions and explore further both mindfulness techniques as needed.
  Interventions: Behavioral: Mindfulness
- Control (No Intervention): Standard of care will be offered to all mothers in the control group which includes kangaroo care but does not involve any mindfulness practices.

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness techniques will be taught to the participants
  Arms: Mindfulness Intervention

SUMMARY:
Very high levels of stress have been reported in parents with their infants admitted to Neonatal Intensive Care Unit (NICU). Review of literature shows that the symptoms are consistent with Post-Traumatic Stress Disorder (PTSD), Acute Stress Disorder and many parents have depression that lasts longer than a month. Skin-to-skin care offers many benefits to the mother and the infant including reduction of maternal stress. However, it has been observed that mothers giving skin-to-skin care for preterm infants in an NICU environment focus on the cardiorespiratory monitoring and its alarms instead of focusing on the baby and "being in the moment". There have also been other challenges noted with maternal sleep while providing skin-to-skin and parental distraction on hand-held devices while providing skin-to-skin. Mindfulness offers a way to focus on being in the moment and accepting the present moment in a non-judgmental and compassionate manner. Mindfulness has been shown to reduce stress in parents of babies admitted to NICU.

To date, they are no studies looking at Mindfulness during skin-to-skin care. This study will explore the feasibility and acceptability of teaching mindfulness skills to mothers providing skin-to-skin care and studying its effects on maternal stress and distraction.

This study involves providing Mindfulness-based strategies during skin-to-skin care to NICU mothers for four consecutive weeks. Participants will be enrolled through informed consent. All participants will be given pre and post participation questionnaires to examine the impact of the sessions on stress reduction, mental wellness and mindfulness quotient. The participants will also be encouraged to maintain a weekly kangaroo care log. Participants will be asked to fill out an acceptability form at the end of the 4 weeks. The data will be analyzed to study the effect of mindfulness on stress reduction and mental wellness. The study will also help understand the uptake and acceptance of such a course by NICU mothers. The results of this study will lead to a future randomized controlled trial looking at the impact of mindfulness practise during skin-to-skin care on parental stress reduction.

DETAILED DESCRIPTION:
BACKGROUND

Kangaroo Mother Care (KMC) was developed to complement neonatal care for premature and low birth weight infants in areas where there were fewer resources. During KMC, a baby is positioned in skin-to-skin contact with the mother's (or father's) chest and each session may last for 30 minutes to a few hours or longer as tolerated. A recent meta-analysis concluded that KMC resulted in better thermal regulation, physiologic stability, enhance breastfeeding and also reduced mortality and infection. KMC has also been shown to improve mother-infant attachment and reduced maternal stress. KMC is widely practiced across the world. Skin-to-Skin care has also been identified with certain challenges and concerns, especially in the immediate neonatal period. There are several instances of the sudden unexpected postnatal collapse of babies reported. In most instances, these episodes were associated with inadequate standardization in selecting mother-baby dyads. There is a strong association with the baby's position, maternal sleep while KMC and inadequate monitoring during KMC. Maternal and neonatal fall while giving KMC has also reported as a concern especially associated with maternal sleep while providing KMC.

KMC in a NICU environment has its own challenges with barriers identified in a recent systematic review including, staffing issues, inadequate training available, difficulties in transferring babies for KMC while attached to infusion pumps and ventilators, stress among caregivers and families. It has also been observed that mothers giving KMC for preterm infants in a NICU environment focus on the cardiorespiratory monitoring and its alarms instead of focusing on the baby and "being in the moment". There have also been other challenges noted with maternal sleep while providing KMC and parental distraction on hand-held devices while providing KMC.

Parents of babies admitted to the NICU undergo a lot of stress. A systematic review of the parental experience of having an infant in the NICU showed that parents experience anxiety and stress. Symptoms of acute stress disorder in 40% of mothers

7-10 days after the birth of the premature infant has been reported in a prospective observational study conducted here at the Stollery Children Hospital, Edmonton. Another study evaluated symptoms of post-traumatic stress disorder (PTSD) and found that 51% of mothers and 33% of fathers screened positive for PTSD.

Mindfulness offers a way to focus on being in the moment and accepting the present moment in a non-judgemental and compassionate manner. Mindfulness has been shown to reduce stress in parents of babies admitted to NICU.

This pilot study is planned to explore the opportunity of teaching Mindfulness skills to mothers providing KMC and studying its effects on maternal stress and distraction. To our knowledge, there are no scientific studies that evaluated mindfulness during kangaroo care or skin-to-skin care.

OBJECTIVE

To explore the feasibility and acceptability of practicing Mindfulness while giving Kangaroo mother care - "Mindful Kangaroo care"

To explore potential benefits of Mindful Kangaroo care, such as stress reduction, change in mindfulness state, variation in screening for depression and anxiety and overall satisfaction with this practice

MATERIALS AND METHODS

This study is a non-blinded, prospective, observational pilot randomized controlled study.

Inclusion and Exclusion Criteria

Postpartum mothers whose baby is receiving care at the Stollery Children Hospital NICU, Royal Alexandra site, are eligible to enter the study.

Mothers would be eligible to participate

a) if they speak, read and write English, b) if their baby is anticipated to require a NICU stay of at least 4 weeks following recruitment, c) if the baby's medical condition allows for skin-to-skin care at recruitment, d) if the mother is available to do regular kangaroo care during the next 4 weeks after recruitment and if the mother is agreeable to receive some teaching for 30-45 minutes weekly during those four weeks.

Mothers whose baby is experiencing imminent risk of death at recruitment will be excluded. Mothers who reported current mental illness issues, current or prior substance abuse/addiction will be excluded.

We aim to recruit 30 participants, 15 in both groups.

Procedure

Once recruited, mothers will be randomized into the mindful kangaroo care intervention group or into the no intervention kangaroo care group. To ensure prior experience with skin-to-skin care, data collection in both groups will begin after the mother has had at least two skin-to-skin experiences with her baby.

Interventions

Mindful Kangaroo Care Group (MKCG)

All research team members are mindfulness practitioners and/or coaches. Some of the researchers would instruct and support weekly, one-on-one, all mothers in their mindfulness practices over a period of 4 weeks.

The MKCG will involve four face-to-face direct coaching on Mindfulness techniques at weekly intervals. The following will be the broad theme of each coaching session

Week 1 - On the first encounter, the mothers will learn how to practice an introductory mindfulness technique to develop the awareness of any sensations felt in the body while holding their baby.

Week 2 - On the second encounter, the mothers will learn how to practice a second mindfulness technique to create positive feelings in the body while holding their baby.

During the third and fourth weekly encounters, the mothers will have a chance to ask their questions and explore further both mindfulness techniques as needed.

Control Group (CG)

Standard of care will be offered to all mothers in the control group which includes kangaroo care but does not involve any mindfulness practices.

The following instruments will be given for the mothers to complete to study the feasibility, acceptability and effect on stress.

Power analysis will not be done because of the pilot study nature; a goal of recruiting a convenience sample of 30 mothers is set. The 30 possible participants will be randomized in a 1:1 ratio (15 participants to each group) at the time of enrollment.

Instruments

* General Demographics Form: A researcher created maternal demographic data form (age, educational level, number of gestations, parity, prior experience with kangaroo care with other children, history of depression/anxiety, gestational age at baby's birth, birth weight, delivery type and infant age at first skin-to-skin experience) to be completed by the mother at enrollment.
* Kangaroo care log: Document recording timing and duration of kangaroo care. Document whether or not the intervention (mindfulness) is practiced using a single-item, 5-point Likert scale (0%, 25%, 50%, 75% or 100% of kangaroo care"). Document how long they used their phones, talk to someone and slept off while doing KMC using the same scale. Document satisfaction with Kangaroo Care for each session using a single-item, 5-point Likert scale ("Very dissatisfied" to "Very satisfied") measuring mother satisfaction with kangaroo care and a space to write any comments. Log to be completed by the mother weekly throughout the study time.
* Mindfulness scale: Toronto Mindfulness Scale as described above to be completed by the mother once at enrollment and at the end of the four weeks. An option will be added to allow the participant to express that she does not understand the statement on the scale.
* Stress scale: Neonatal Unit Parental Stressor Scale as described above, to be completed by the mother once at enrollment and at the end of the four weeks.
* Depression and Anxiety scale: Patient Health Questionnaire 4, as described above, to be completed by the mother once at enrollment and at the end of the four weeks.
* Feasibility form: A researcher created a data form to evaluate the recruitment capability, the data collection procedures and outcome measures, the resources and ability to manage and implement the study and intervention, to be completed by the investigators throughout the study time.
* Acceptability form: A researcher created a 3-point Likert scale ("unacceptable" to "acceptable") measuring mother acceptability to the different instruments (demographic form and the outcome scales) and acceptability to the intervention, to be completed by the mother at the end of the four weeks.

Statistical analyses

Descriptive statistics will be calculated to summarize sample characteristics and will be compared between groups. Appropriate statistical tests (independent and paired t-tests, Wilcoxon signed-rank test, Mann-Whitney U tests and χ2 tests) will be used to examine for differences between study group demographics, for differences between groups independent study variables (parent stress score, mindfulness score), and for within-group changes in both scores from before to after the intervention. Given our small sample size, we are primarily interested in exploring the direction of any effects. Feasibility data will be analyzed by descriptive statistics where appropriate and qualitatively where appropriate. Acceptability data will be evaluated using descriptive statistics.

Possible Risks:

The risk is minimal. Mindfulness practice trains the brain to develop attention skills. There might be challenges that may arise during mindfulness meditation. Those challenges are usually the same that arise during normal daily life. When they occur during mindfulness, they become opportunities to develop insight. Should a mother had an overwhelming experience, the people offering mindfulness instructions to her would be able to help her. Moreover, the social workers on our unit are trained to respond to acute distress, they are aware of this research project and are willing to support the mothers as needed.

Possible Benefits:

There may or may not be a direct benefit to the mothers from taking part in this study. Some people experience less stress, less anxiety, less intrusive thoughts, less confusion or less foggy mind with a mindfulness practice. Some people experience more satisfaction, more fulfilment, or they become more aware of their emotions, more aware of their thinking process, more presence in their interactions and relationships. The information that we will gather may improve the care of other mothers.

ELIGIBILITY:
Inclusion Criteria:

* Mothers would be eligible to participate

  1. if they speak, read and write English,
  2. if their baby is anticipated to require a NICU stay of at least 4 weeks following recruitment,
  3. if the baby's medical condition allows for skin-to-skin care at recruitment,
  4. if the mother is available to do regular kangaroo care during the next 4 weeks after recruitment and
  5. if the mother is agreeable to receive some teaching for 30-45 minutes weekly during those four weeks.

Exclusion Criteria:

* Mothers whose baby is experiencing imminent risk of death at recruitment will be excluded.
* Mothers who reported current mental illness issues, current or prior substance abuse/addiction will be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in stress symptoms | Change from recruitment to 4 weeks after
  Using the Parental Stressor Scale for NICU parents. Parents rate the amount of stress. Scores for each question range from 1 (not at all stressful) to 5 (extremely stressful). A higher score indicates a higher level of stress.
Change in anxiety symptoms | Change from recruitment to 4 weeks after
  Using the Patient Health Questionnaire 4. Scores for each question range from 1 (not at all) to 4 (nearly every day). A higher score suggests anxiety.
Change in depression symptoms | Change from recruitment to 4 weeks after
  Using the Patient Health Questionnaire 4. Scores for each question range from 1 (not at all) to 4 (nearly every day). A higher score suggests depression.
Acceptability | 4 weeks after recruitment
  A researcher created 3-point Likert scale, measuring acceptability of the different instruments and mindfulness intervention during the research project

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Antoine Landry, MD, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, NICU, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No